CLINICAL TRIAL: NCT05138835
Title: A Randomized, Double Blind Evaluation of the Effects of BOTOX® Cosmetic on Skin Health
Brief Title: BOTOX® Cosmetic and Skin Health.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andreas Nikolis (Other)
Responsible Party: Sponsor-Investigator, Andreas Nikolis, Medical Director, Erevna Innovations Inc.
Organization: Erevna Innovations Inc. (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-ALG-BTX
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Oily Skin
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Subjects will receive BTX in the glabella and forehead regions, using a traditional injection technique commonly utilized in aesthetic medicine. The traditional injection technique will deposit the neurotoxin into the targeted muscles; with up to 24 units being injected into the forehead and 20 units in the glabella.
  Interventions: Drug: Botox Cosmetic
- Group 2 (Experimental): Subjects will receive the traditional, deep injection technique, in addition to a superficial intradermal injection technique, which uses micro-aliquots of toxin. The superficial technique will deposit 0.1 units of toxin at 5mm intervals, at the level of the deep dermis.
  Interventions: Drug: Botox Cosmetic

INTERVENTIONS:
Drug: Botox Cosmetic — BOTOX® Cosmetic is approved and commercially available for use in Canada.
  BOTOX® Cosmetic is a prescription medicine that is injected into muscles and used to temporarily improve the look of moderate to severe frown lines between the eyebrows, crow's feet lines, and forehead lines in adults.

SUMMARY:
This is a two cohort, randomized, double blind, single center study to evaluate the effects of Botox Cosmetic (BTX) on sebum protection. Thirty-four female subjects with moderate-to-high skin sebum concentration will be recruited and randomized in a 1:1 ratio to treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years.
2. Female sex.
3. A SebumeterTM score >66ug/cm2 at Baseline.
4. Ability to adequately understand the verbal explanations and the written subject information provided in local language and ability and willingness to give consent to participate in the study.
5. Signed and dated informed consent to participate in the study and unrestricted use of facial images for marketing purpose.
6. If female of childbearing potential: a negative urine pregnancy test before all treatments is required.
7. Subject agrees to use the same topical cosmetic products (e.g., cleansers, moisturizers) throughout the duration of the trial, and at least for 30 days prior to enrolment.
8. Subject is on a stable diet and is not planning any major dietary changes throughout the duration of the trial.
9. Subject is not planning on undergoing any major hormonal changes throughout the duration of the study (e.g., menopause, change in medications).

Exclusion Criteria:

1. Current Pregnancy or lactation [sexually active women of childbearing age must agree to use medically acceptable methods of contraception for the duration of this study (e.g., oral contraceptives, condoms, intrauterine device, shot/injection, patch)];
2. Patients meeting any official BOTOX® Cosmetic contra-indications;
3. Inability to comply with follow-up and abstain from other treatments in the region of interest during the study period;
4. Heavy smokers, classified as smoking more than 12 cigarettes per day;
5. History of severe or multiple allergies manifested by anaphylaxis;
6. Previous tissue revitalization therapy in the treatment area within 6 months before treatment with laser or light, mesotherapy, radiofrequency, ultrasound, cryotherapy, chemical peeling, or dermabrasion;
7. Previous treatment with neurotoxins in the area under assessment, within 6 months prior to enrolment;
8. Previous treatment with soft tissue fillers in the area under assessment, within 6 months prior to enrolment;
9. Subjects presenting with known allergy to BOTOX® Cosmetic.
10. Subjects presenting with porphyria.
11. Subjects with active disease, such as inflammation, infection or tumors, in or near the intended treatment site.
12. History of bleeding disorders or treatment with thrombolytics, anticoagulants, or inhibitors of platelet aggregation (e.g. Aspirin or other non-steroid anti-inflammatory drugs [NSAIDs]), within 2 weeks before treatment.
13. Subjects using immunosuppressants.
14. Subjects prescribed systematic or topical (in the area under assessment) antibiotics within 1 month of enrolment.
15. Tattoos, piercings or visible markings that in the treating investigator's opinion, may interfere with results or assessments.
16. Cancer or precancer in the treatment area, e.g. actinic keratosis.
17. Patients with a tendency to form hypertrophic scars or any other healing disorders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-12-11 (Actual)

PRIMARY OUTCOMES:
Skin quality assessment | Baseline versus Week 4
  Reduction in sebum

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Nikolis, Principal Investigator — Erevna Innovations Inc.
Locations (1):
- Erevna Innovations Inc, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No